CLINICAL TRIAL: NCT02158637
Title: Validation Study of the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-002504 / MC1091; MC1091 (Other: Mayo Clinic)
Record Dates: First submitted 2014-06-04; First posted 2014-06-09 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: PRO-CTCAE; Patient-Reported Outcomes; Common Terminology Criteria for Adverse Events; Questionnaire; Adverse Events; Symptoms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients receiving treatment: Patients receiving active treatment for cancer or initiating treatment for cancer in the next 7 days

SUMMARY:
This study is being done to try out questions from a large set of questions called the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). The PRO-CTCAE is a set of questions which asks patients about their symptoms. This study will look at properties of these questions and will provide information about how these questions can be improved for research studies. PRO-CTCAE questions were developed under a contract from the National Cancer Institute (NCI) to allow patients to self-report symptoms in future cancer clinical trials. Patients with cancer receiving treatment will complete a web-based questionnaire containing PRO-CTCAE questions and a paper booklet containing a commonly used questionnaire for assessing quality of life, functioning, and symptoms at two visits one to six weeks apart. Some patients will additionally complete web-based questionnaires containing PRO-CTCAE questions weekly for four to five weeks, while completing a daily questionnaire containing PRO-CTCAE questions using an automated telephone system. Lastly, a small number of patients will complete only a single visit in which a web-based, telephone-based, and paper-based questionnaire containing PRO-CTCAE items is completed in addition to a paper booklet containing a commonly used questionnaire for assessing quality of life, functioning, and symptoms. The primary hypothesis is that scores for PRO-CTCAE questions will differ between patients with high versus low general well-being as measured by your doctor using a scale called the Eastern Cooperative Oncology Group Performance Score.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Disease and treatment matching 1 of 7 following cohorts: breast cancer receiving chemotherapy or initiating chemotherapy in the next 7 days; lymphoma/myeloma receiving chemotherapy or initiating chemotherapy in the next 7 days; metastatic prostate or bladder cancer receiving chemotherapy or initiating chemotherapy in the next 7 days; metastatic or locally advanced lung cancer receiving chemotherapy or initiating chemotherapy in the next 7 days or receiving radiation therapy for greater than or equal to 21 more days; metastatic colorectal cancer receiving chemotherapy or initiating chemotherapy in the next 7 days; head, neck, or gastroesophageal cancer receiving radiation therapy for greater than or equal to 21 more days; any cancer enrolled through an National Cancer Institute Community Cancer Centers Program site
* Willing to return to registering institution in 1-6 weeks (subset only)
* Eastern Cooperative Oncology Group Performance Status 0-4
* Ability to understand English and read questions on a computer screen
* Ability to hear and respond to questions in English using a telephone keypad (subset only)
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Willing to be reached at a single telephone number (without extension or operator involvement) for the next 21 to 28 days (subset only)
* Ability to participate in the study visit lasting 45-60 minutes total, including the informed consent process, being shown by study staff how to use each mode of administration (computer, automated telephone, and paper), and completing questionnaires (subset only)

Exclusion Criteria:

* Clinically significant cognitive or memory impairment in the opinion of clinical or research staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients initiating or receiving chemotherapy, radiation therapy, or both at nine U.S.-based cancer centers and community oncology practices were approached in clinical waiting areas and invited to participate in this questionnaire-based study.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
Difference in PRO-CTCAE item scores between patients with good and poor performance status at the first visit (study day 1) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Amylou C. Dueck, PhD, Study Chair — Mayo Clinic
Locations (9):
- United States (9):
  - St. Joseph Hospital of Orange, Orange, California
  - Hartford Hospital, Hartford, Connecticut
  - Christiana Care Health Services, Wilmington, Delaware
  - The Cancer Program of Our Lady of the Lake and Mary Bird Perkins, Baton Rouge, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer, New York, New York
  - Gibbs Cancer Center, Spartanburg, South Carolina
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Lee MK, Mitchell SA, Basch E, Deal AM, Langlais BT, Thanarajasingam G, Ginos BF, Rogak L, Mendoza TR, Bennett AV, Noble BN, Mazza GL, Dueck AC. Psychometric Properties and Interpretability of PRO-CTCAE(R) Average Composite Scores as a Summary Metric of Symptomatic Adverse Event Burden. Cancers (Basel). 2025 Oct 28;17(21):3459. doi: 10.3390/cancers17213459. PMID 41228252
- [Derived] Lee MK, Mitchell SA, Basch E, Mazza GL, Langlais BT, Thanarajasingam G, Ginos BF, Rogak L, Meek EA, Jansen J, Deal AM, Carr P, Blinder VS, Jonsson M, Mody GN, Mendoza TR, Bennett AV, Schrag D, Dueck AC. Identification of meaningful individual-level change thresholds for worsening on the patient-reported outcomes version of the common terminology criteria for adverse events (PRO-CTCAE(R)). Qual Life Res. 2025 Feb;34(2):495-507. doi: 10.1007/s11136-024-03819-5. Epub 2024 Nov 6. PMID 39503942
- [Derived] Bennett AV, Dueck AC, Mitchell SA, Mendoza TR, Reeve BB, Atkinson TM, Castro KM, Denicoff A, Rogak LJ, Harness JK, Bearden JD, Bryant D, Siegel RD, Schrag D, Basch E; National Cancer Institute PRO-CTCAE Study Group. Mode equivalence and acceptability of tablet computer-, interactive voice response system-, and paper-based administration of the U.S. National Cancer Institute's Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). Health Qual Life Outcomes. 2016 Feb 19;14:24. doi: 10.1186/s12955-016-0426-6. PMID 26892667